CLINICAL TRIAL: NCT07247383
Title: A Phase II, Prospective Clinical Trail to Evaluate the Efficacy and Safety of Orelabrutinib Combined With Low-Dose Radiotherapy or Rituximab in the Treatment of Ocular Adnexal MALT Lymphoma
Brief Title: Orelabrutinib Plus Low-Dose Radiotherapy Or Rituximab For Ocular Adnexal MALT Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0995
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Marginal Zone Lymphoma of Ocular Adnexal; Marginal Zone Lymphoma(MZL)
Keywords: Marginal zone lymphoma; Orelabrutinib; Phase II Trail: Orelabrutinib Plus Low-Dose Radiotherapy Or Rituximab For Ocular Adnexal MALT Lymphoma（Efficacy & Safety）
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; Radiotherapy; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AnnArbor 1 (Experimental): Radiotherapy 2GY * 2 + Orelabrutinib 150 mg qd; 28 days per cycle for 4 cycles
  Interventions: Drug: Orelabrutinib (ICP-022); Radiation: radiotherapy
- AnnArbor 2 (Experimental): Rituximab plus Orelabrutinib 150 mg QD, 28 days per cycle for 4 cycles
  Interventions: Drug: Orelabrutinib (ICP-022); Drug: Rituximab (R)
- AnnArbor 3-4 (Experimental): Rituximab plus Orelabrutinib 150 mg QD, 28 days per cycle for 6 cycles
  Interventions: Drug: Orelabrutinib (ICP-022); Drug: Rituximab (R)

INTERVENTIONS:
Drug: Orelabrutinib (ICP-022) — Orelabrutinib was administered in 4 or 6 cycles, respectively, based on subjects' AnnArbor stage as assessed by PETCT，150mg QD D1-28
Radiation: radiotherapy — Radiotherapy 2Gy*2
  Arms: AnnArbor 1
Drug: Rituximab (R) — Rituximab 375mg/m2 D1
  Arms: AnnArbor 2; AnnArbor 3-4

SUMMARY:
This is a phase II, prospective clinical study to evaluate the efficacy and safety of Orelabrutinib combined with Low-Dose Radiotherapy or Rituximab in the treatment of Ocular Adnexal MALT Lymphoma

DETAILED DESCRIPTION:
Marginal zone lymphoma (MZL) is a relatively common type of B-cell non-Hodgkin's lymphoma (B-NHL), with an incidence rate second only to diffuse large B-cell lymphoma (DLBCL) and follicular lymphoma (FL). According to different clinical manifestations and pathological features, it is divided into three subtypes: mucosa-associated lymphoid tissue lymphoma (MALT), also known as extranodal marginal zone lymphoma, nodal marginal zone lymphoma (NMZL), and splenic marginal zone lymphoma (SMZL). The incidence of MZL increases with age. The median age at diagnosis for EMZL patients is 60 years old. Its characteristics are mainly indolent, and most are limited to the site of origin. The 5-year overall survival rate and 10-year overall survival rate are 88.7% and 81.4%, respectively; the median overall survival period is 13 years. The median age at diagnosis for SMZL patients is 65 years old. Its characteristics are mainly indolent, and 25-30% of patients show aggressive behavior. The 5-year overall survival rate and 10-year overall survival rate are 79.7% and 57.9%, respectively; the median overall survival period is 9 years (aggressive < 4 years). The median age at diagnosis for NMZL patients is usually between 50 and 60 years old. Its characteristics are usually aggressive. The 5-year overall survival rate and 10-year overall survival rate are 76.5% and 62.8%, respectively; the median overall survival period is 8 years. Although the overall survival period of MZL is long, patients often relapse and may face multiple relapses. Therefore, choosing an appropriate treatment strategy for MZL is particularly important.

Among them, mucosa-associated lymphoid tissue extranodal marginal zone (MALT) lymphoma is a low-grade non-Hodgkin's lymphoma derived from B cells. Its clinical course is relatively indolent and it often occurs in mucosa-associated lymphoid tissues of extranodal organs. Orbital adnexal lymphoma (OAL) is the most common malignant tumor of the orbital adnexa in adults, accounting for 1% to 2% of all lymphomas and 8% of extranodal lymphomas. MALT lymphoma is the most common pathological type of OAL. Orbital adnexal MALT lymphoma (OAML) accounts for 80% to 98% of OAL in Asia and 50% to 78% in Western countries. OAML is MALT lymphoma that involves the orbital adnexa (eyelids, conjunctiva, lacrimal glands, orbit, etc.). In China, the incidence is higher in men than in women, with a median age of 45 to 60 years. Most lesions only invade the local and surrounding tissues of the orbital adnexa, and some patients have lymph node or distant organ involvement. The clinical manifestations are damage to the morphology and function of the involved organs, with a slow disease course. Most patients have a good prognosis.

Most OAML lesions are limited to the orbital adnexa, with the most frequently involved site being the orbit (>40%), followed by the conjunctiva (35% to 40%), eyelids (10% to 15%), and lacrimal glands (≤10%). When local lesions are extensive, composite lesions may occur, that is, multiple sites of the orbital adnexa are involved at the same time; a small number of patients have involvement of tissues and organs outside the orbital adnexa. Unilateral involvement is more common, but a few also present with bilateral involvement. Most patients do not have B symptoms such as fever, weight loss, and night sweats. Pathological examination is the gold standard for lymphoma diagnosis. Due to the lack of obvious specific manifestations in the clinical manifestations and imaging examinations of OAML, this disease must be diagnosed through pathological examination.

A real-world study of OAML included 694 OAML patients from 11 centers in China. Among them, 229 patients received a watch-and-wait (W&W) strategy after diagnosis of OAML due to no residual lymphoma lesions or symptoms after surgery. A total of 160 cases (34.4%) received radiotherapy (RT) with a dose of 24 to 36 Grays. 187 cases (40.2%) received immunotherapy and chemotherapy regimens such as R-CHOP, R-CVP, BR, or CHOP, CVP, etc. 11 patients received rituximab treatment. 8 patients received a combination of rituximab and local ocular radiotherapy. The best response was evaluated for 455 patients who received postoperative consolidation therapy. The overall response rate (ORR) was 94.5% (including 237 cases of complete response and 193 cases of partial response), and 5 patients had disease progression. The median follow-up was 731 days (12-7443), and a total of 142 patients had disease progression or recurrence (20.5%), including 130 cases of intraocular recurrence and 12 cases (8.5%) of extraocular recurrence. Only 1 patient was defined as histological transformation to DLBCL. 47 patients received salvage RT treatment, of which 45 achieved remission (95.7%), including 23 cases of complete remission. 18 patients died, and only 3 patients died of lymphoma-related events. The 10-year overall survival rate was 95.5%, and the 10-year lymphoma-specific overall survival rate was 99.3%. Adverse events in patients receiving RT included dry eye syndrome in 33 cases (20.6%), vision loss in 16 cases (10%), and cataracts in 2 cases (1.3%). This indicates that the safety of RT for OAML still needs to be further improved. The 2025 NCCN guidelines also point out that for the eye area, a low dose should be selected first, and 4 Gy in two fractions can be used as an alternative to 24 Gy. When using this extremely low-dose regimen, it is crucial to have regular and careful follow-up with radiation oncologists and ophthalmologists (including appropriate physical examinations and imaging studies). For patients with incomplete remission or recurrence, a definitive dose is recommended.

BTK belongs to the non-receptor tyrosine protein TEC family and is expressed in B lymphocytes, mast cells, macrophages, monocytes, neutrophils, etc. It is a key molecule in B cell antigen receptor (BCR) signaling and controls B cell development and differentiation by activating cell cycle positive regulators and differentiation cytokines. It also controls B cell survival and proliferation by regulating the expression of pro-apoptotic and anti-apoptotic proteins. BTK inhibitors target the BCR signaling pathway to inhibit B cell maturation and activation.

The preliminary exploration results of BTKi in first-line MZL are encouraging. Acalabrutinib, as a new-generation BTK inhibitor, has high selectivity compared to other BTK inhibitors. Previous studies have shown that at a concentration of 1 µM, it inhibits more than 90% of BTK among 456 tested kinases, making it the BTK inhibitor with the highest kinase selectivity reported so far. The adverse reactions are mainly headache, fatigue, etc., mostly mild, and the overall tolerance is good. Based on the results of the phase II clinical trial of acalabrutinib in treating marginal zone lymphoma, on April 21, 2023, the new BTK (Bruton's tyrosine kinase) inhibitor acalabrutinib was approved by the National Medical Products Administration (NMPA) of China for the treatment of relapsed/refractory marginal zone lymphoma (MZL) patients, becoming the first and currently the only small molecule targeted drug with MZL indication in China. The study showed that for patients with relapsed/refractory MZL who had received at least one treatment including CD20 monoclonal antibodies, the ORR of acalabrutinib monotherapy was 57.8%, the CRR was 12%, and the median DOR was 34.3 months. A study explored the efficacy and safety of orelabrutinib combined with ultra-low-dose radiotherapy in the treatment of ocular adnexal extranodal marginal zone B-cell lymphoma. A total of 21 patients with OA-EMZL were included, among which 3 patients had bilateral involvement and the remaining 18 patients had unilateral involvement. 17 patients completed the treatment, with an ORR of 100% (17/17) and a CR rate of 94.1% (16/17). During orelabrutinib treatment, 8 patients did not experience early toxic reactions such as dermatitis, dry eye, conjunctivitis, or lacrimation. One patient who had undergone lacrimal gland resection did not experience aggravated dry eye symptoms. The combination of ultra-low-dose radiotherapy and orelabrutinib for OAML not only improved the treatment effect but also significantly reduced the toxic reactions of radiotherapy, providing a new treatment option for localized OAML.

Although radiotherapy is widely used in OAML and has achieved significant efficacy, it still has some shortcomings. For example, the traditional radiotherapy dose is relatively high, which may lead to a series of ocular complications such as cataracts, dry eye, and keratitis. These complications not only affect the visual function of patients but also have a significant negative impact on their quality of life. In addition, the long-term side effects of radiotherapy may gradually emerge several years after treatment, increasing the long-term follow-up and management burden of patients. Therefore, exploring more efficient and low-toxicity treatment options for OAML patients is a valuable scientific and clinical attempt. For this reason, this study explored the combination of orelabrutinib with low-dose radiotherapy and orelabrutinib with CD20 monoclonal antibody rituximab in the treatment of OAML, in order to provide more comprehensive and effective treatment options for OAML patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged ≥18 years, with no gender restriction;
* 2. Patients with OAML confirmed by histopathology;
* 3. Ann Arbor stage (I~II);
* 4. ECOG performance status score of 0-2;
* 5. No previous systemic treatment;
* 6. Major organ functions meet the following criteria:
* (1). Blood routine: Absolute neutrophil count ≥1.5×10⁹/L, platelet count ≥75×10⁹/L, hemoglobin ≥75g/L; In case of bone marrow involvement, absolute neutrophil count ≥1.0×10⁹/L, platelet count ≥50×10⁹/L, hemoglobin ≥50g/L;
* (2). Blood biochemistry: Total bilirubin ≤1.5×ULN, AST or ALT ≤2×ULN; Serum creatinine ≤1.5×ULN; Serum amylase ≤ULN;
* (3). Coagulation function: International Normalized Ratio (INR) ≤1.5×ULN.
* 7. Expected survival time ≥3 months
* 8. Voluntarily sign a written informed consent form before trial screening.

Exclusion Criteria:

* 1. Current or previous history of other malignant tumors, except those with evidence of no recurrence or metastasis for at least 5 years after radical treatment;
* 2. Lymphoma involving the central nervous system or transformed to high-grade lymphoma;
* 3. Non-hematological toxicities from previous anti-tumor treatment have not recovered to ≤ Grade 1 (except alopecia);
* 4. Uncontrolled or significant cardiovascular diseases, including:
* (1). Congestive heart failure of New York Heart Association (NYHA) Class II or higher, unstable angina pectoris, myocardial infarction within 6 months before the first administration of the study drug, or arrhythmia requiring treatment at screening, or left ventricular ejection fraction (LVEF) < 50%;
* (2). Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, unclassified cardiomyopathy);
* (3). History of clinically significant QTc interval prolongation, or QTc interval at screening (female > 470ms, male > 450ms);
* (4). Subjects with symptomatic coronary heart disease requiring medication;
* (5). Subjects with poorly controlled hypertension (blood pressure not reaching the target after more than 1 month of using 3 or more reasonable and tolerable maximum-dose antihypertensive drugs (including diuretics) on the basis of lifestyle modification, or blood pressure can only be effectively controlled by taking 4 or more antihypertensive drugs);
* 5. Active bleeding within 2 months before screening, or current use of anticoagulant drugs, or clear bleeding tendency as judged by the investigator;
* 6. Urine protein ≥ 2+, and 24-hour urine protein quantification ≥ 2g/24h;
* 7. History of deep vein thrombosis or pulmonary embolism within 6 months before screening;
* 8. History of organ transplantation or allogeneic bone marrow transplantation;
* 9. Major surgery performed within 6 weeks before screening or minor surgery performed within 2 weeks before screening. Major surgery refers to surgery requiring general anesthesia, while endoscopic examination for diagnostic purposes is not considered major surgery. Insertion of vascular access devices is exempted from this exclusion criterion;
* 10. Active infection, or uncontrolled HBV (HBsAg positive and/or HBcAb positive with positive HBV DNA titer), HCV Ab positive, HIV/AIDS, or other severe infectious diseases;
* 11. Subjects with severe pulmonary function impairment such as current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, etc.;
* 12. Previous treatment with BTK inhibitors, BCR pathway inhibitors (e.g., PI3K, Syk) and BCL-2 inhibitors;
* 13. Eligible for and planning to undergo stem cell transplantation;
* 14. Any mental or cognitive impairment that may limit the understanding and execution of the informed consent form and compliance with the study;
* 15. Subjects with drug addiction or alcoholism;
* 16. Pregnant or lactating women, and fertile subjects who are unwilling to take contraceptive measures;
* 17. Continuous use of drugs with moderate-to-severe inhibitory or strong inductive effects on cytochrome P450 CYP3A;
* 18. Other conditions deemed unsuitable for participating in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CR) | up to 6 months
  The rate of patients who achieved complete response after treatment

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 6 months
  ORR is defined as the proportion of patients with a response of CR or PR
Progression free survival (PFS) | Up to 2 years
  The time from when a patient starts treatment to when the disease progresses or the patient dies for any reason.
Overall Survival | Up to 2 years
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
Adverse Event (AE) | After signing the ICF until 28 Days (± 7 days) after the last dose
  Any adverse medical event that occurred between the time the patient signed informed consent and the end of the trial was an adverse event, regardless of whether it was causally related to the trial drug.

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No